CLINICAL TRIAL: NCT00116740
Title: A 12-Week, Dose-Ranging, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of APD356 in Obese Patients
Brief Title: Safety and Efficacy of APD356 in the Treatment of Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-004
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2006-12

CONDITIONS: Obesity
Keywords: Serotonin; 5-HT2c; Satiety; Obesity; Appetite suppressant; Weight Loss; Overweight
MeSH Terms: conditions — Obesity; Anorexia; Weight Loss; Overweight | interventions — lorcaserin

INTERVENTIONS:
Drug: APD356

SUMMARY:
This is a research study of an investigational drug, APD356, a novel, selective 5-HT2c receptor agonist, in clinical development as a potential treatment for obesity.

The purpose of this study is to obtain a preliminary assessment of the safety and efficacy of APD356, when administered daily for 12 weeks, in obese subjects who are otherwise healthy. Subjects who are on concomitant medications for control of hypertension or blood lipids may qualify.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, parallel group study. Three different doses of APD356 or placebo will be administered daily for 12 weeks, to obese, male and nonpregnant, nonlactating, female volunteers, aged 18 to 65 years. Approximately 400 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or nonpregnant, nonlactating females aged 18-65 years (inclusive)
* Body mass index (BMI) of 30-45 kg/m2
* Non-smoker
* No concomitant medications other than hypertension medications (stable > 90 days) and/or statins (stable > 90 days)
* No past treatment with drugs associated with the development of pulmonary hypertension or cardiac valvular insufficiency
* No more than mild mitral valve regurgitation and absence of aortic valve regurgitation upon screening echocardiogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-06; Study Completion 2005-11

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Safety
Changes in waist circumference, hip circumference, and waist/hip ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Smith SR, Prosser WA, Donahue DJ, Morgan ME, Anderson CM, Shanahan WR; APD356-004 Study Group. Lorcaserin (APD356), a selective 5-HT(2C) agonist, reduces body weight in obese men and women. Obesity (Silver Spring). 2009 Mar;17(3):494-503. doi: 10.1038/oby.2008.537. Epub 2008 Dec 4. PMID 19057523
- See also: obesity information — http://www.obesityonline.org/
- See also: N. American Association for the Study of Obesity web page — http://www.obesity.org/
- See also: sponsor company web page — http://www.arenapharm.com
- See also: Pennington Biomedical Research Center home web page — http://www.pbrc.edu